CLINICAL TRIAL: NCT05266352
Title: Investigation of the Effect of Exercise Training on Psychosocial Outcomes in Rotator Cuff
Brief Title: Investigation of the Effect of Exercise Training on Psychosocial Outcomes in Rotator Cuff Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 108
Record Dates: First submitted 2022-02-28; First posted 2022-03-04 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-03

CONDITIONS: Rotator Cuff Tears; Pain, Shoulder; Psychological
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supervised exercise group (Experimental): The group received the supervised exercise program
  Interventions: Other: Supervised exercise program
- Home exercise group (Active Comparator): The group received the home exercise program
  Interventions: Diagnostic Test: Home exercise program

INTERVENTIONS:
Other: Supervised exercise program — A structured program consisting of range of motion, postural control, scapulothoracic strengthening, glenohumeral strengthening and dynamic stabilization exercises used in conservative treatment of rotator cuff tears will be performed for 8 weeks.
  Patients will do the exercises under control of the physiotherapist in the clinic.
  Arms: Supervised exercise group
Diagnostic Test: Home exercise program — A structured program consisting of range of motion, postural control, scapulothoracic strengthening, glenohumeral strengthening and dynamic stabilization exercises used in conservative treatment of rotator cuff tears will be performed for 8 weeks.
  Patients will do the exercises at home. Patients will visit the clinic every 2 weeks and progression of exercise program will be made.
  Arms: Home exercise group

SUMMARY:
This study aimed to determine the psychosocial effects of exercise training in patients with rotator cuff tears.

DETAILED DESCRIPTION:
This study aimed to determine the psychosocial effects of exercise training in patients with rotator cuff tears. Fifty voluntary patients with partial rotator cuff tear will be randomized into two groups: Supervised exercise group (SE) and home exercise (HE) group, for a standardized 8 weeks exercise program. The primary outcome is the Constant-Murley Score (CMS). The secondary outcomes are the Visual Analogue Scale (VAS), active range of motion (AROM), Pain Catastrophizing Scale (PCS), Hospital Anxiety and Depression Scale (HADS), Pittsburgh Sleep Quality Index (PSI), Short Form-12 (SF-12), and Global Rating of Change (GRC). Outcome measures will be performed at baseline and at the end of 8-week intervention.

ELIGIBILITY:
Inclusion Criteria: Forty years of age or older patients that have been diagnosed for a partial rotator cuff tear that is unrelated to trauma by a specialist orthopedist with MRI and physical examination and no other shoulder problems on the diagnosed shoulder will be included into this study.

Exclusion Criteria: Patients diagnosed with full-thickness or massive rotator cuff tear, patients who undergone previous surgery, patients diagnosed with frozen shoulder or glenohumeral instability, and athletic patients younger than 40 years of age with symptoms of acute RC tear will not be included into this study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Constant-Murley Score | Baseline
  The functional level will be assessed by the Constant Murley Score, which is a 100-point scale consisting of 15 points for pain, 20 points for daily activities, 40 points for pain-free range of motion, and 25 points for strength. High scores are positively correlated with the increased functional level. While pain and activities of daily living are evaluated by the patient, range of motion and strength are evaluated by the clinician.

SECONDARY OUTCOMES:
Constant-Murley Score | At the end of 8-week intervention
  The functional level will be assessed by the Constant Murley Score, which is a 100-point scale consisting of 15 points for pain, 20 points for daily activities, 40 points for pain-free range of motion, and 25 points for strength. High scores are positively correlated with the increased functional level. While pain and activities of daily living are evaluated by the patient, range of motion and strength are evaluated by the clinician.
Visual Analogue Scale (VAS) | Baseline
  Pain intensity will be measured using the visual analogue scale (VAS). The participants will be asked to indicate their perceived pain at rest, during activity and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on 10 cm line using a ruler. The higher scores indicate an higher level of pain.
Visual Analogue Scale (VAS) | At the end of 8-week intervention
  Pain intensity will be measured using the visual analogue scale (VAS). The participants will be asked to indicate their perceived pain at rest, during activity and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on 10 cm line using a ruler. The higher scores indicate an higher level of pain.
Active Range of Motion (AROM) Assessment | Baseline
  The shoulder flexion, abduction, internal and external rotation ROM will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a digital goniometer. The process will be repeated three times in each direction, with the average value recorded.
Active Range of Motion (AROM) Assessment | At the end of 8-week intervention
  The shoulder flexion, abduction, internal and external rotation ROM will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a digital goniometer. The process will be repeated three times in each direction, with the average value recorded.
Pain Catastrophizing Scale (PCS) | Baseline
  Pain catastrophizing, which is characterized by the tendency to magnify the threat value of a pain stimulus and to feel helpless in the presence of pain, as well as by a relative inability to prevent or inhibit pain-related thoughts in anticipation of, during, or following a painful event will be measured using the Pain Catastrophizing Scale (PCS).
Pain Catastrophizing Scale (PCS) | At the end of the 8-week intervention
  Pain catastrophizing, which is characterized by the tendency to magnify the threat value of a pain stimulus and to feel helpless in the presence of pain, as well as by a relative inability to prevent or inhibit pain-related thoughts in anticipation of, during, or following a painful event will be measured using the Pain Catastrophizing Scale (PCS).
The Hospital Anxiety and Depression Scale (HADS) | Baseline
  The anxiety and depression will be assessed using the Pain Catastrophizing Scale (PCS), which is used to measure anxiety and depression in a general medical population of patients.
The Hospital Anxiety and Depression Scale (HADS) | At the end of the 8-week intervention
  The anxiety and depression will be assessed using the Pain Catastrophizing Scale (PCS), which is used to measure anxiety and depression in a general medical population of patients.
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  The anxiety and depression will be assessed using the Pittsburgh Sleep Quality Index (PSQI), which is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval.
Pittsburgh Sleep Quality Index (PSQI) | At the end of the 8-week intervention
  The anxiety and depression will be assessed using the Pittsburgh Sleep Quality Index (PSQI), which is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval.
Short Form-12 (SF-12) | Baseline
  Health related quality of life will be assessed using the SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
Short Form-12 (SF-12) | At the end of the 8-week intervention
  Health related quality of life will be assessed using the SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
Global Rating of Change (GRC) | At the end of the 8-week intervention
  Patient satisfaction regarding improvement in shoulder function will be assessed by the Global Rating of Change (GRC) scale. The patients will be asked to rate their condition after a 8-week intervention period compared to baseline by indicating whether they have improved significantly, improved slightly, unchanged, deteriorated slightly, or deteriorated significantly in this study.
Exercise Dairy | At the end of the 8-week intervention
  A self reported adherence to home exercise program will be assessed using the exercise dairy.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, PT, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)